CLINICAL TRIAL: NCT06342141
Title: Empagliflozin for Reducing the Risk of No-Reflow Phenomenon in Patients Undergoing Percutaneous Coronary Intervention for ST-Elevation Myocardial Infarction
Brief Title: Empagliflozin for No-reflow Phenomenon in PCI for STEMI
Acronym: EMPA-PCI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto Nacional de Cardiologia Ignacio Chavez (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 24-1423
Record Dates: First submitted 2024-03-11; First posted 2024-04-02 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2024-07

CONDITIONS: STEMI; No-Reflow Phenomenon
MeSH Terms: conditions — ST Elevation Myocardial Infarction; No-Reflow Phenomenon | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Empagliflozin (Experimental): The patients included in this group will receive a loading dose of 25 mg of Empagliflozin at the time of enrollment in the study, prior to percutaneous coronary intervention. Over the following three days, they will receive a daily maintenance dose of 10 mg of Empagliflozin.
  Interventions: Drug: Empagliflozin 25 milgrams (Mg); Drug: Empagliflozin 10 Mg
- Standar Treatment (No Intervention): The patients included in this group will receive standar treatment according to the current guidelines

INTERVENTIONS:
Drug: Empagliflozin 25 milgrams (Mg) — Load dose
  Other Names: Jardiance 25 Mg
  Arms: Empagliflozin
Drug: Empagliflozin 10 Mg — Maintenance dose
  Other Names: Jardiance 10 Mg
  Arms: Empagliflozin

SUMMARY:
Myocardial infarction remains, in our current era, a leading cause of morbidity and mortality both domestically and globally. A significant contributor to this issue is reperfusion injury, which enlarges the infarction, deteriorates ventricular function, leads to poorer outcomes, and currently has no specific treatment. Originally developed as an antidiabetic, empagliflozin has shown significant benefits in other organs and systems. Recent years have seen the demonstration of its cellular and vascular effects in animal models, potentially contributing to the reduction of reperfusion damage. However, no human studies have yet confirmed these effects.

Consequently, this randomized, parallel-arm clinical trial was designed to evaluate the effect of empagliflozin treatment, administered from the pre-intervention period through to 3 days post-intervention, on the incidence of the no-reflow phenomenon in patients with ST-segment elevation myocardial infarction (STEMI) undergoing coronary angioplasty compared to a placebo.

Before entering the hemodynamics room, participants in the intervention group will receive a loading dose of 25 mg of empagliflozin or a standar treatment. In-hospital treatment will continue with 10 mg empagliflozin daily for 3 days for the intervention group. Patients will be monitored weekly during the first month and bi-weekly during the second and third months.

The primary outcome will be the incidence of the no-reflow phenomenon, measured through the Thrombolysis in Myocardial infarction (TIMI) flow scale in the coronary angiography performed to treat the infarction. Secondary outcomes will include the reduction of ST segment on the electrocardiogram, troponin levels, differences in the longitudinal strain by echocardiogram, and infarct size by magnetic resonance imaging.

ELIGIBILITY:
Inclusion Criteria:

* Acute myocardial infarction with ST-segment elevation
* Presentation to the institute within 12 hours of symptom onset
* Coronary angioplasty chosen as the reperfusion treatment for the subject
* Known diagnosis of diabetes or admission glucose >180 mg/dl.
* Informed consent signed

Exclusion Criteria:

* Hemodynamically unstable subjects
* Subjects undergoing thrombolysis treatment in the current event
* History of coronary revascularization surgery
* Known allergy or hypersensitivity to Sodium-glucose co-transporter-2 (SGLT2) inhibitors
* History of recurrent urinary tract infections
* Known chronic kidney disease and estimated glomerular filtration rate (eGFR) < 20
* Ongoing treatment with any SGLT2 inhibitor
* Participation in another clinical trial or having participated in the week prior to recruitment
* For women of childbearing age: Current or planned pregnancy or lactation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2024-08-22 (Actual); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Non-Reflow Phenomenon | During percutaneous coronary intervention (approximately 60 minutes after receiving the loading dose)
  Incidence of non-reflow phenomenon during percutaneous coronary intervention measured using the Thrombolysis in myocardial infarction (TIMI) Flow Grading System. Dichotomous variable (yes/no).
  The TIMI flow grading system ranges from 0 to 3. Grade 3 flow is the best result of angioplasty and means that flow has been restored to normal. Grade 2 flow means that the contrast flows throughout the entire artery but more slowly than normal. Grade 1 flow means that the contrast flows through the artery but does not reach the end of the artery. Flow grade 0 means that contrast does not flow in the artery. It is the worst result of an angiography. Any flow other than grade 3 is interpreted as a non-reflow phenomenon.

SECONDARY OUTCOMES:
Infract size | 72 hours after the loading dose
  Myocardial infarct size measured in grams using cardiac magnetic resonance. Continuous variable. Mean difference between both groups. This outcome will not be combined with other secondary outcomes.
Longitudinal Strain | 24 hours after the loading dose
  Longitudinal Strain measured in percentage using transthoracic echocardiogram. Continuous variable. Mean difference between both groups. This outcome will not be combined with other secondary outcomes.
High-sensitivity Troponin Clearance | 72 hours after the loading dose
  Percentage of High-sensitivity troponin decrease when comparing admission values with values at 72 hours. Continuous variable. Mean difference between both groups. This outcome will not be combined with other secondary outcomes.
Creatine Kinase-myocardial band Clearance | 72 hours after the loading dose
  Percentage of creatine kinase-myocardial band (CK-MB) decrease when comparing admission values with values at 72 hours. Continuous variable. Mean difference between both groups. This outcome will not be combined with other secondary outcomes.
Adverse Cardiovascular Events | Up to 3 months after the loading dose
  Incidence of Rehospitalization, malignant arrhythmias, cardiogenic shock, reinfarction, urgent revascularization, death. This outcome will not be combined with other secondary outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Arias-Sanchez, MD, Principal Investigator — Deputy Head of the Department of Interventional Cardiology at the National Institute of Cardiology
Locations (1):
- National Institute of Cardiology, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Niccoli G, Kharbanda RK, Crea F, Banning AP. No-reflow: again prevention is better than treatment. Eur Heart J. 2010 Oct;31(20):2449-55. doi: 10.1093/eurheartj/ehq299. Epub 2010 Sep 13. No abstract available. PMID 20837571
- [Background] Tasar O, Karabay AK, Oduncu V, Kirma C. Predictors and outcomes of no-reflow phenomenon in patients with acute ST-segment elevation myocardial infarction undergoing primary percutaneous coronary intervention. Coron Artery Dis. 2019 Jun;30(4):270-276. doi: 10.1097/MCA.0000000000000726. PMID 31026233
- [Background] Niccoli G, Burzotta F, Galiuto L, Crea F. Myocardial no-reflow in humans. J Am Coll Cardiol. 2009 Jul 21;54(4):281-92. doi: 10.1016/j.jacc.2009.03.054. PMID 19608025
- [Background] Annibali G, Scrocca I, Aranzulla TC, Meliga E, Maiellaro F, Musumeci G. "No-Reflow" Phenomenon: A Contemporary Review. J Clin Med. 2022 Apr 16;11(8):2233. doi: 10.3390/jcm11082233. PMID 35456326
- [Background] Sayour AA, Korkmaz-Icoz S, Loganathan S, Ruppert M, Sayour VN, Olah A, Benke K, Brune M, Benko R, Horvath EM, Karck M, Merkely B, Radovits T, Szabo G. Acute canagliflozin treatment protects against in vivo myocardial ischemia-reperfusion injury in non-diabetic male rats and enhances endothelium-dependent vasorelaxation. J Transl Med. 2019 Apr 16;17(1):127. doi: 10.1186/s12967-019-1881-8. PMID 30992077
- [Background] Cooper S, Teoh H, Campeau MA, Verma S, Leask RL. Empagliflozin restores the integrity of the endothelial glycocalyx in vitro. Mol Cell Biochem. 2019 Sep;459(1-2):121-130. doi: 10.1007/s11010-019-03555-2. Epub 2019 May 24. PMID 31127491
- [Background] Lahnwong C, Palee S, Apaijai N, Sriwichaiin S, Kerdphoo S, Jaiwongkam T, Chattipakorn SC, Chattipakorn N. Acute dapagliflozin administration exerts cardioprotective effects in rats with cardiac ischemia/reperfusion injury. Cardiovasc Diabetol. 2020 Jun 15;19(1):91. doi: 10.1186/s12933-020-01066-9. PMID 32539724
- [Background] Shao Q, Meng L, Lee S, Tse G, Gong M, Zhang Z, Zhao J, Zhao Y, Li G, Liu T. Empagliflozin, a sodium glucose co-transporter-2 inhibitor, alleviates atrial remodeling and improves mitochondrial function in high-fat diet/streptozotocin-induced diabetic rats. Cardiovasc Diabetol. 2019 Nov 28;18(1):165. doi: 10.1186/s12933-019-0964-4. PMID 31779619
- [Background] Kolijn D, Pabel S, Tian Y, Lodi M, Herwig M, Carrizzo A, Zhazykbayeva S, Kovacs A, Fulop GA, Falcao-Pires I, Reusch PH, Linthout SV, Papp Z, van Heerebeek L, Vecchione C, Maier LS, Ciccarelli M, Tschope C, Mugge A, Bagi Z, Sossalla S, Hamdani N. Empagliflozin improves endothelial and cardiomyocyte function in human heart failure with preserved ejection fraction via reduced pro-inflammatory-oxidative pathways and protein kinase Galpha oxidation. Cardiovasc Res. 2021 Jan 21;117(2):495-507. doi: 10.1093/cvr/cvaa123. PMID 32396609
- [Background] Lu Q, Liu J, Li X, Sun X, Zhang J, Ren D, Tong N, Li J. Empagliflozin attenuates ischemia and reperfusion injury through LKB1/AMPK signaling pathway. Mol Cell Endocrinol. 2020 Feb 5;501:110642. doi: 10.1016/j.mce.2019.110642. Epub 2019 Nov 21. PMID 31759100
- [Background] Tan Y, Yu K, Liang L, Liu Y, Song F, Ge Q, Fang X, Yu T, Huang Z, Jiang L, Wang P. Sodium-Glucose Co-Transporter 2 Inhibition With Empagliflozin Improves Cardiac Function After Cardiac Arrest in Rats by Enhancing Mitochondrial Energy Metabolism. Front Pharmacol. 2021 Oct 12;12:758080. doi: 10.3389/fphar.2021.758080. eCollection 2021. PMID 34712142
- [Background] Uthman L, Li X, Baartscheer A, Schumacher CA, Baumgart P, Hermanides J, Preckel B, Hollmann MW, Coronel R, Zuurbier CJ, Weber NC. Empagliflozin reduces oxidative stress through inhibition of the novel inflammation/NHE/[Na+]c/ROS-pathway in human endothelial cells. Biomed Pharmacother. 2022 Feb;146:112515. doi: 10.1016/j.biopha.2021.112515. Epub 2021 Dec 9. PMID 34896968
- [Background] Seo MS, Jung HS, An JR, Kang M, Heo R, Li H, Han ET, Yang SR, Cho EH, Bae YM, Park WS. Empagliflozin dilates the rabbit aorta by activating PKG and voltage-dependent K+ channels. Toxicol Appl Pharmacol. 2020 Sep 15;403:115153. doi: 10.1016/j.taap.2020.115153. Epub 2020 Jul 24. PMID 32717242
- [Background] Zou R, Shi W, Qiu J, Zhou N, Du N, Zhou H, Chen X, Ma L. Empagliflozin attenuates cardiac microvascular ischemia/reperfusion injury through improving mitochondrial homeostasis. Cardiovasc Diabetol. 2022 Jun 15;21(1):106. doi: 10.1186/s12933-022-01532-6. PMID 35705980
- [Derived] Solis-Jimenez F, Araiza-Garaygordobil D, Masso-Bueso JS, Villalobos-Ordaz A, Arellano-Juvera F, Arredondo-Aragon F, Melendez-Ramirez G, Valdez-Ortiz R, Alday-Ramirez SM, Rodriguez-Zanella HG, Amezcua Guerra LM, Arias-Mendoza MA, Martinez-Rios MA, Arias-Sanchez EA, Eid-Lidt G. Effect of empagliflozin on reducing the no-reflow phenomenon in patients with ST-elevation myocardial infarction: rationale and design of the EMPA-PCI trial. Eur Heart J Open. 2025 Oct 5;5(6):oeaf128. doi: 10.1093/ehjopen/oeaf128. eCollection 2025 Nov. PMID 41230400